CLINICAL TRIAL: NCT06857409
Title: The Effect of Suprascapular Nerve Pulsed Radiofrequency Treatment on Central Sensitization and Neuropathic Pain
Brief Title: Suprascapular Nerve PRF for Central Sensitization and Neuropathic Pain
Acronym: SSPRF-CS
Status: Active, not recruiting | Type: Observational
Sponsor: Gülçin Babaoğlu (Other)
Responsible Party: Sponsor-Investigator, Gülçin Babaoğlu, Medical doctor, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Other Study IDs: TABED 2-25-949
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-02

CONDITIONS: Shoulder Pain
Keywords: shoulder pain; suprascapular nerve; radiofrequency; central sensitization; neuropatic pain
MeSH Terms: conditions — Shoulder Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suprascapular nerve pulsed radiofrequency: patients undergoing suprascapular nerve pulsed radiofrequency therapy
  Interventions: Procedure: pulsed radiofrequency

INTERVENTIONS:
Procedure: pulsed radiofrequency — All patients will be monitored with electrocardiography, non-invasive blood pressure, and peripheral oxygen saturation, and peripheral intravenous vascular access will be performed before the procedure. Patients will be placed in a sitting position. The physician will stand behind the patient for the posterior approach. The skin area to be injected will be prepared and covered in a sterile manner using a povidone-iodine-based solution. The operator will use ultrasound (a TOSHIBA Aplio 500 Ultrasound) guidance to perform suprascapular nerve radiofrequency. The suprascapular notch will be visualized. A twenty-two gauge, 10 cm long, and 10 mm active-tipped radiofrequency cannula will be introduced to the suprascapular notch. Motor stimulation will be performed at 2 Hz at a setting of 1 V, and sensory stimulation will be performed at 50 Hz at a setting of 0.5 V. After the needle tip confirmation, pulsed radiofrequency will be applied to the suprascapular nerve for 360 seconds.

SUMMARY:
Chronic shoulder pain affects quality of life and is often associated with central sensitization, leading to treatment resistance. Pulsed radiofrequency (PRF) of the suprascapular nerve, which innervates 70% of the shoulder joint, is a promising therapy for nociceptive and neuropathic pain. This study evaluates the effects of PRF on central sensitization and neuropathic pain in chronic shoulder pain. Clinical assessments will be conducted at baseline, 1 month, and 3 months post-treatment to determine PRF's potential in reducing central sensitization and improving shoulder function.

DETAILED DESCRIPTION:
Chronic shoulder pain is a prevalent musculoskeletal condition affecting quality of life, with an incidence of 18-26% in the general population. Its prevalence has doubled over the past 40 years. Pain sensitization, independent of etiology, is frequently observed in patients with musculoskeletal shoulder pain and can lead to poorer clinical outcomes even after primary disease treatment. Chronic pain development involves both peripheral and central sensitization mechanisms, with central sensitization characterized by amplified pain signaling and reduced inhibitory pathway activity. This can result in pain persistence independent of tissue damage and resistance to treatment.

Conventional treatments for chronic shoulder pain include physiotherapy, nonsteroidal anti-inflammatory drugs (NSAIDs), and intra-articular steroid injections. However, these may not provide sufficient long-term analgesia, and some patients develop treatment-resistant chronic pain. Recently, pulsed radiofrequency (PRF) treatment applied to the suprascapular nerve, responsible for 70% of the sensory innervation of the shoulder joint, has gained attention for its efficacy in reducing both nociceptive and neuropathic pain. PRF modulates neural activity without causing thermal damage and may have the potential to reduce central sensitization. However, its effects on central sensitization and neuropathic pain mechanisms remain insufficiently studied.

This study aims to evaluate the impact of suprascapular nerve PRF on central sensitization and neuropathic pain in chronic shoulder pain. Clinical assessments will be conducted at baseline, 1 month, and 3 months post-treatment to examine changes in central sensitization, neuropathic pain, and shoulder function. This study seeks to determine whether PRF can serve as an effective alternative in chronic shoulder pain management by reducing central sensitization and improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Chronic shoulder pain persisting for at least 3 months
* Radiologically confirmed shoulder lesions, including:

Rotator cuff tendinopathy Adhesive capsulitis Bursitis Osteoarthritis

* At least two positive provocation tests (Neer, Hawkins, Jobe tests)
* Shoulder pain resistant to conservative treatments, including:

Nonsteroidal anti-inflammatory drugs (NSAIDs) Physical therapy Corticosteroid injections

Exclusion Criteria:

* Traumatic shoulder pain (e.g., fractures, dislocations)
* History of shoulder surgery
* Active inflammation or rheumatic diseases affecting the shoulder, including:

Rheumatoid arthritis Polymyalgia rheumatica Ankylosing spondylitis

* Cervical radiculopathy
* Central nervous system diseases, such as:

Multiple sclerosis Stroke Spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic shoulder pain persisting for at least 3 months
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory (CSI) | baseline, 1st and 3rd months
  The CSI will be used to assess symptoms related to CS. The CSI will consist of two parts, Part A and Part B. Part A will include 25 items scored on a scale from 0 to 100, with higher scores indicating an increased CS-related symptom burden. In Part B, diagnoses of central sensitivity syndromes will be questioned, and this part will not be included in the scoring.

SECONDARY OUTCOMES:
Douleur Neuropathique 4 (DN4) Questionnaire | baseline, 1st and 3rd months
  The DN4 questionnaire is a screening tool used to identify neuropathic pain. It consists of 10 items, with seven related to sensory symptoms (burning, painful cold, electric shocks, tingling, pins and needles, numbness, and itching) and three based on a clinical examination (hypoesthesia to touch, hypoesthesia to pinprick, and pain triggered by brushing). Each item is scored as 1 (present) or 0 (absent), with a total score ranging from 0 to 10.
Numerical Rating Scale (NRS) | baseline, 1st and 3rd months
  The Numerical Rating Scale (NRS) is a widely used pain assessment tool that allows patients to rate their pain intensity on a scale from 0 to 10, where:
  0 = No pain 10 = Worst imaginable pain
Shoulder Pain and Disability Index (SPADI) | baseline, 1st and 3rd months
  The Shoulder Pain and Disability Index (SPADI) is a self-reported questionnaire designed to assess pain and functional impairment in individuals with shoulder disorders. It consists of 13 items divided into two subscales:
  Pain Subscale (5 items) - Evaluates the intensity of shoulder pain during different activities.
  Disability Subscale (8 items) - Assesses the difficulty in performing daily activities due to shoulder problems.
  Each item is scored on a numerical scale from 0 to 10, with 0 = no pain or difficulty and 10 = worst pain or extreme difficulty. The total score ranges from 0 to 100, with higher scores indicating greater pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: ERKAN YAVUZ AKÇABOY, Prof. Dr., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided